CLINICAL TRIAL: NCT01928797
Title: To Determine if the Cardiac Output Monitoring During Cesarean Delivery Under Spinal Anesthesia Will Change Our Clinical Practice of Using Vasopressors
Brief Title: Ninvasive Cardiac Output Measurements During Cesarean Delivery Under Spinal Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bhavani Shankar Kodali, Vice Chair, Anesthesiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-p-001314
Record Dates: First submitted 2012-10-02; First posted 2013-08-27 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Hypotension During Cesarean Delivery; Spinal Anesthesia
Keywords: cardiac output pregnancy spinal anesthesia

STUDY DESIGN:
Intervention Model Description: Investigator randomly assigns the subjects into one of the two groups. Control group and Interventional group
Masking Description: The investigator assigned the subject to one of the groups. Care provided followed the protocol for the group and the investigator analyzed the outcome results.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The care provider will use blood pressure and heart rate data to administer vasopressor use. In the control group, vasopressors (phenylephrine and ephedrine) will be used as considered appropriate to maintain BP within 20% of baseline. The CO data is measured and blinded to the anesthesiologists in the control group, therefore the anesthesiologist choice of ephedrine or phenylephrine is based on the individual anesthesiologist standard of care preference
- Study group (Experimental): The care provider will use the cardiac output monitor data (intervention) to guide vasopressors (Phenylephrine and ephedrine) in addition to blood pressure and heart rate data based on a standardized protocol in addition to the blood pressure and heart rate data available in the control group.
  Interventions: Device: Cardiac output monitor data

INTERVENTIONS:
Device: Cardiac output monitor data — The availability of cardiac output monitor provides additional hemodynamic indices that may help guide anesthesiologists to better select vasopressors
  Arms: Study group

SUMMARY:
The purpose of the study is to learn more about how the heart works during cesarean delivery under spinal anesthesia (medicines given in the spine that numb parts of your body to block pain) in women. The investigators would like to find out if the information about the heart can help in treating blood pressure changes that occur during the cesarean delivery. The investigators would also like to find out if this information can help reduce the chances of nausea and vomiting during the cesarean delivery.

The activity of the heart changes during spinal anesthesia and cesarean section. In the past, a sensor placed directly into the heart was the only way to see how the heart worked. Currently, there are monitors that can sense the heart's activity via sensors that are placed on the skin during cesarean delivery.

In this study, the investigators will use the ICON cardiac output (ICON) monitor. The ICON monitor is approved by the US Food and Drug Administration (FDA) to monitor (check) the activity of your heart.

This study aims to:

1. Determine if additional cardiac output measurements help anesthesiologists maintain appropriate hemodynamics as defined as within 20% of baseline BP and if it changed their choice of vasopressors (primary outcome).
2. Determine if additional cardiac output measurements help to decrease the incidence of nausea and vomiting during cesarean delivery (secondary outcome).

DETAILED DESCRIPTION:
Most women who undergo elective cesarean delivery in our hospital have spinal anesthesia for the surgery. You will receive standard spinal anesthesia techniques whether or not you take part in this study. You will be asked to sign a separate clinical consent form for the spinal anesthesia and for your cesarean delivery.

After the anesthesiologist places your spinal anesthesia, the investigator will record your blood pressure every two minutes as is the standard practice in our institution. An anesthesiologist is a doctor who specializes in giving drugs or other agents to prevent or relieve pain during surgery or other procedures. The investigator will also continuously record your heart rate and the amount of oxygen in your blood as is the standard practice. If needed, the anesthesiologist will give you medications to maintain your blood pressure.

In addition to the standard procedures described above, additional monitoring (checking) of your heart will be performed as part of this study. The investigator will use the ICON monitor to measure the amount of blood pumped by each heart beat.

The anesthesiologist will put on the sensors (sticky pads). There are four sticky pads that are similar to what is used during electrocardiograms (EKGs). Two sensors are placed on the left side of your neck and two on the left side of your trunk. The sensors have wires attached that will be plugged into a small heart monitor device that records the information.

The investigators will place the sensors on you before you receive the spinal anesthesia. The sensors will record what your heart is doing before placement of spinal anesthesia until the end of your surgery.

The investigators will assign you by chance (like a coin toss) to one of the following groups:

* Group Study: Your anesthesiologist will have access to the amount of blood that is pumped during each heart beat. The anesthesiologist will treat and maintain the amount of blood pumped during each beat so that it is within the normal range.
* Group Control: Your anesthesiologist will NOT have access to the amount of blood that is pumped during each heart beat. The anesthesiologist will treat and maintain your blood pressure throughout your delivery. (This is the current routine care.)

The control group and the study group will receive spinal anesthesia as is adapted in our institution. HR and BP will be measured every two minutes as is normal practice. Cardiac output will be measured in all patients in both groups. The subjects will have four surface ECG electrodes attached to the left side of the neck and the lower thorax (at the level of the xiphoid). Baseline hemodynamic parameters (SV (stroke volume), HR (heart rate), CO (cardiac output) , SVV (stroke volume variation), and SVR (systemic vascular resistance)) will be determined before placing spinal anesthesia. Continuous CO data will be recorded by the unit.

In the study group, phenylephrine and ephedrine will be used depending on the blood pressure and cardiac output data. If the CO is normal, and BP is below 20% of baseline, phenylephrine boluses of 40 micrograms at two minute interval (BP recording time) will be used to maintain BP within 20% of the baseline. If the BP is normal, but CO is lower than 20% baseline, ephedrine boluses (10 mg) will be used. If BP and CO is lower, a combination of both phenylephrine and ephedrine will be used.

In the control group, the phenylephrine and ephedrine will be used as considered appropriate to maintain BP within 20% of baseline. The CO data will be blinded to the anesthesiologists in the control group

Study group (algorithm in detail):

1. If SBP<20%, CO is within (<,± ) 20% of baseline: Phenylephrine 40 mic boluses to bring BP within 20% of the baseline.
2. If CO < 20%, and BP is within (<,± ) 20% of baseline, ephedrine boluses to bring the CO.
3. If both are below 20% of baseline, phenylephrine 40 mic boluses and ephedrine 10 mg together will be used at 2 min intervals until both reach to within 20% of baseline.
4. If SBP is normal, and CO is greater than 20% baseline, no treatment needed.
5. If CO is normal, and SBP is greater than 20%, no treatment needed.

Control group:

Although BP and CO are being measured in the control group, CO data is blinded to the clinician. Therefore the clinician will use SPB data and current practice instincts to choose either of vasopressors considered appropriate to treat hypotension.

The anesthesiologist has his or her discretion of treating BP, or CO if these parameters are not corrected with above protocol.

Fluid inputs and outputs will be noted that includes blood loss. Apgar scores of newborns will be obtained from neonatologists' assessment. Incidence of nausea and vomiting and medications used will be also noted.

The regional techniques will follow the standards adopted by our institution. Most placements are done in the sitting position. After disinfecting the skin with betadine in the usual fashion, the patients back will be draped with a sterile clear plastic and local anesthetic (1.5 % lidocaine, 2ml) injected at the site of placement. A 3 1/2 -inch 25-gauge Whittaker needle will be inserted into the spinal space at either the L3-L4 or L4-L5. Once the clear Cerebrospinal fluid (CSF) is obtained, spinal medication (1.6 - 1.8 ml of bupivacaine 0.75% with hyperbaric dextrose, 10 µgm fentanyl, 200 µgm morphine). Most patients receive oxytocin infusion titrated to uterine tone (3-5 units/hr) and ondansetron for prevention of postoperative nausea and vomiting after delivery of the baby.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant subjects

Exclusion Criteria:

* Other than healthy
* High blood pressure. Presumed excessive bleeding, medications for blood pressure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11-01; Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Shankar Kodali, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start Date: November 2013 Types of location: Brigham and Women's Hospital Labor and Delivery Unit
Groups:
- Control Group: Vasopressor use based on blood pressure and heart rate. Cardiac output data was blinded to the care providers.
- Study Group: Vasopressor use based on the cardiac output, blood pressure and heart rate.
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: cardiac output monitor will be attached CO values will not be used to guide vasopressor use. The care provider will use blood pressure and heart rate data to guide vasopressor use.
- Study Group: cardiac output monitor will be attached CO values will guide vasopressor use in addition blood pressure and heart rate
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (5.6) | 34.3 (5.3) | 34.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Cardiac Output [Mean (Standard Deviation); unit: L/min] | 6.3 (1.3) | 6.5 (1.3) | 6.4 (74)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Cardiac Output Within and Outside 20% of Baseline Values
Description: To determine mean cardiac output differences between the control group and the study group that used cardiac output data. In the control group, the cardiac output data was measured but not used for correcting blood pressure changes. Blood pressure changes were used for administering phenylephrine or ephedrine. In the study group, cardiac output data was used, in addition to blood pressure data, to correct both cardiac output and blood pressures to be maintained within 20% of baseline measurements.
  After spinal anesthesia for cesarean delivery, the cardiac output and blood pressure tends to decrease. When this occurs, the blood flow to the uterus and the baby decrease resulting in fetal heart changes. Since we do not monitor the baby during the actual cesarean delivery (technically difficult), the strategy is to maintain the blood pressure and cardiac output within the 20% of the baseline values.
Time Frame: intraoperatively during surgery
Measure: Number; unit: percentage of patients
Groups:
- Control Group: cardiac output monitor will be attached but CO values will not guide vasopressor use as CO data is blinded to care provider
- Study Group: cardiac output monitor will be attached and CO data used to guide management based on the protocol
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
percentage of patients
  Percent incidences (CO within 20% baseline) | 71 | 66
  Percent incidences (CO outside 20% baseline | 29 | 34
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.37, Chi-squared

2. Secondary Outcome: Nausea and Vomiting
Description: incidence of nausea, and vomiting
Time Frame: intraoperatively during surgery
Population: Nausea
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Vasopressor use based on the blood pressure changes and heart rate
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants
  Incidence of vomiting | 1 | 1
  Incidence of Nausea | 9 | 9
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.33, Chi-squared

3. Secondary Outcome: Number of Participants With Umbilical Cord pH
Description: Number of participants with Umbilical cord pH <7.2
Time Frame: Intraoperative
Population: 1 out of 30 babies had umbilical pH < 7.2
Measure: Number; unit: number of participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
number of participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Intraoperative period
Groups:
- Control Group: cardiac output monitor will be attached but will not guide treatment based on cardiac output. The treatment will be based on blood pressure changes.
- Study Group: cardiac output monitor will be attached CO values will guide vasopressor protocol use
Arm/Group | Control Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=30) | Study Group (N=30)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No